CLINICAL TRIAL: NCT05170451
Title: A Randomized Controlled Trial of Topical Cannabidiol for the Treatment of Musculoskeletal Pain
Brief Title: Topical CBD for Musculoskeletal Pain
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Terminated due to hurdles of obtaining regulatory approval.
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Brent DeGeorge, Assistant Professor of Plastic Surgery, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSR200170
Record Dates: First submitted 2021-12-10; First posted 2021-12-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Musculoskeletal Pain
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with crossover
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Comparator: Start with CBD (Active Comparator): The study design with be a double-blind, randomized controlled trial with crossover. Treatment will be blinded to the subjects and investigators. Patients will be randomly assigned 2 weeks of the CBD and then crossover to the other condition (Shea butter only) for 2 additional weeks. Patients will apply the topical cream to the affected body region or joint two times daily for 1 hour. Subjects will be advised to observe for physiologic changes, skin changes, or other adverse effects.
  Interventions: Drug: CBD; Other: Control
- Active Comparator: Start with control (Shea butter) (Active Comparator): The study design with be a double-blind, randomized controlled trial with crossover. Treatment will be blinded to the subjects and investigators. Patients will be randomly assigned 2 weeks of Shea butter and then crossover to the other condition (CBD) for 2 additional weeks. Patients will apply the topical cream to the affected body region or joint two times daily for 1 hour. Subjects will be advised to observe for physiologic changes, skin changes, or other adverse effects.
  Interventions: Drug: CBD; Other: Control

INTERVENTIONS:
Drug: CBD — Topical CBD 50 mg/ml applied in 1mL amounts twice daily
Other: Control — Topical shea butter applied in 1mL amounts twice daily
  Other Names: Shea butter

SUMMARY:
Rationale: CBD is commonly being used as an over-the-counter treatment for musculoskeletal pain; however, no clinical trial has been performed to establish efficacy of CBD in humans for musculoskeletal pain.

Hypothesis: CBD is more effective than placebo for relieving pain and improving patient-reported outcomes for musculoskeletal pain.

Study Design: The study design with be a double-blind, randomized controlled trial with crossover. Treatment will be blinded to the subjects and investigators. Patients will be randomly assigned 2 weeks of the CBD or control and then crossover to the other condition for 2 additional weeks. Patients will apply the CBD or control cream to the affected area twice daily (approximately every 12 hours) for 1 hour. Subjects will be advised to observe for physiologic changes, skin changes, or other adverse effects.

DETAILED DESCRIPTION:
Study Population: 100 subjects presenting with musculoskeletal pain over the age of 18 will be recruited from the University of Virginia from the Hand Center or Primary Care Clinic.

Description of Sites/Facilities Enrolling Participants: This will be a single-site study conducted at the University of Virginia in the Hand Center and the Primary Care Clinic.

Description of Study Intervention: The study design will be a double-blind randomized control trial with crossover. Treatment will be blinded to the subjects and investigators. Patients will be randomly assigned 2 weeks of the case (CBD) or control cream and then crossover to the other cream for 2 more weeks with a 1-week washout interval between. Patients will apply the topical cream to the affected body region or joint two times daily for 1 hour. The subjects will be advised to observe for physiologic changes, skin changes, or other adverse effects. If mild to severe adverse events are noticed, the creams will be removed immediately, and appropriate care and observation will be taken. Each condition will last for 2 weeks and then subjects will be contacted by the study coordinator to facilitate crossover into the other condition following a 1-week washout period. To capture any delayed-onset adverse events, including those related to skin changes that might develop after the drug is discontinued, subjects will attend a follow-up visit seven days following the last dose of investigational cream.

Study Duration: This study will last one year from the beginning of subject recruitment to data analysis.

Participant Duration: Subjects will be enrolled in this study for approximately seven (7) weeks from Screening until the final Study Visit.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male or female, aged 18 years or older.
4. Females of childbearing potential must have a negative urine and blood pregnancy test at Screening and a negative urine pregnancy test before study drug is administered. Females must abstain from sex or use a highly effective method of contraception during the period from Screening to administration of study drug and for 30 days after the last dose of study medication. Standard acceptable methods include abstinence or the use of a highly effective method of contraception, including; hormonal contraception, diaphragm, cervical cap, vaginal sponge, condom with spermicide, vasectomy, intrauterine device. If females are of non-child bearing potential, they must be post-menopausal defined as: age > 55 with no menses within the past 12 months, or history of hysterectomy, or history of bilateral oophorectomy, or bilateral tubal ligation.
5. Males must consent to use a medically acceptable method of contraception throughout the entire study period and for 90 days after their last study drug application. They must agree to not donate sperm for 90 days after their last study drug application.
6. Presence of physician-diagnosed musculoskeletal pain in a discrete body region, including bone or joint-related pain, tendon or ligament-related pain, muscle-related pain, or fibromyalgia or physician-diagnosed postoperative pain in a discrete body region.

Exclusion Criteria:

1. Subject does not speak English.
2. Subject is blind.
3. Severe cardiac, pulmonary, liver and /or renal disease.
4. Coumadin use at time of screening.
5. History of mental illness.
6. Subjects who are incarcerated.
7. History of drug or substance abuse.
8. Pre-existing CBD or hemp-based product usage.
9. Subject has had a corticosteroid injection ≤ 3 months prior.
10. Subject has had prior surgery for osteoarthritis treatment.
11. Females who are pregnant, nursing or planning a pregnancy; females of childbearing potential who are unwilling or unable to use an acceptable method of contraception as outlined in this protocol from Screening to the first dose of study medication and for 30 days after the last dose of study medication. Standard acceptable methods include abstinence or the use of a highly effective method of contraception, including; hormonal contraception, diaphragm, cervical cap, vaginal sponge, condom with spermicide, vasectomy, intrauterine device.
12. Any skin disease or condition, including eczema, psoriasis, melanoma, acne or contact dermatitis, scarring, imperfections, lesions, tattoos or discoloration that may affect treatment application, application site assessments, or affect absorption of the study drug.
13. Subjects with ALT/AST >3 times the upper limit of normal at screening.
14. Subjects with history of or active depression or suicide ideation based on Columbia-Suicide Severity Rating Scale (C-SSRS).
15. Subjects taking prescription or non-prescription medication which are substrates of CYP3A4 (Itraconazole, Ketoconazole, Azamulin, Troleandomycin, Verapamil, John's wart, Phenobarbital), CYP2C19 (Nootkatone, Ticlopidine, Rifampin, Omeprazole), CYP2C8 (Montelukast, Quercetin, Phenelzine, Rifampin, Clopidogrel) , CYP2C9 (Sulfaphenazole, Tienilic acid, Carbamazepine, Apalutamide, Fluconazole, Celecoxib), CYP1A2 (alpha-Naphthoflavone, Furafylline, Phenytoin, Rifampin, Ritonavir, smoking, Teriflunomide, Ciproflaoxacin, oral contraceptives, Alloprinol) and CYP2B6 (Sertraline, Phencyclidine, Thiotepa, Ticlopidine, Carbamazepine, Efavirenez, Rifampin, Bupropion) within 14 days of the study procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with change in The PROMIS-29 (Patient-Reported Outcomes Measurement Information System) during intervention and at follow-up. | [Time Frame: Every 1 week during intervention and 1 week washout, up to 7 weeks.]
  PROMIS-29 will measure health-related quality of life and is a validated, 29 question survey divided into seven sub-domains of function including physical functioning, social function, pain interference, pain intensity, sleep, depression, and anxiety, where a higher score indicates more pain interference.
Change from baseline in Visual Analog Pain (VAS) Score during intervention and at follow-up. | [Time Frame: Every 1 week during intervention and 1 week washout, up to 7 weeks.]
  The VAS score is a unidimensional measure of pain intensity and is a validated, subjective measure for acute and chronic pain. A patient is asked to indicate his/her perceived pain intensity along a horizontal line (from 0 to 100), and this rating is then measured from the left edge with higher numbers indicating more pain.
Change from baseline in Single Assessment Numerical Evaluation (SANE) | [Time Frame: Every 1 week during intervention and 1 week washout, up to 7 weeks.]
  The SANE score is a validated metric for musculoskeletal pain which can be applied to any joint or region of interest. The patient is asked to rate his/her pain from 0-100. Patients rate their current illness score in relation to their pre-injury baseline.

SECONDARY OUTCOMES:
Rate of side effects using novel CBD cream. | [Time Frame: Daily during intervention and 1 week washout, up to 7 weeks.]
  Side effects will be assessed at each encounter clinical evaluation by patient report in a Symptom Diary. All side effects thought to be secondary to CBD will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Brent DeGeorge, MD, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No